CLINICAL TRIAL: NCT06093100
Title: Wearable Technology to Evaluate Hyperglycemia and Heart Rate Variability in Duchenne Muscular Dystrophy
Brief Title: Wearable Technology to Evaluate Hyperglycemia and HRV in DMD - Longitudinal Aim
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jaclyn Tamaroff, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: 231407
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; heart failure; cardiomyopathy; hyperglycemia; heart rate variability
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Heart Failure; Cardiomyopathies; Hyperglycemia | interventions — Wearable Electronic Devices; Exercise Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: wearable technology — Three wearable devices
  Other Names: Continuous glucose monitor (CGM): The Dexcom G6 Pro Continuous Glucose Monitoring System (Dexcom G6 Pro System); Holter Monitor: Body Guardian Mini Remote Monitoring System; Physical activity and sleep monitor: ActiGraph GT9X accelerometers

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is an X-linked disorder that causes muscle wasting, cardiopulmonary failure, and premature death. Heart failure is a leading cause of death in DMD, but substantial knowledge gaps exist regarding predisposing risk factors. In the general population, hyperglycemia, insulin resistance, and decreased heart rate variability (HRV; reflecting autonomic dysfunction) are associated with cardiomyopathy (CM). It is unclear whether these factors are associated with DMD-CM. Closing this knowledge gap may lead to novel screening and therapeutic strategies to delay progression of DMD related CM. Despite risk factors for hyperglycemia, including the use of glucocorticoids, low muscle mass, obesity, and reduced ambulation, little is known regarding glucose abnormalities in DMD. Some of these same risk factors, along with the distance needed to travel for specialty care, present significant barriers to research participation and clinical care for individuals with DMD. Remote wearable technology may improve research participation in this vulnerable population. Therefore, this study will leverage remote wearable technologies to overcome these barriers and define the relationship between dysglycemia and DMD-CM.

In this Aim of the study, the investigators will assess the utility of remote wearable technology to predict changes in traditional metrics of metabolism and cardiac function. In this pilot study, 10 individuals with DMD will undergo cardiac magnetic resonance imaging (CMR) and oral glucose tolerance tests (OGTTs) at baseline and two years. The investigators will remotely assess glycemia (using continuous glucose monitors), HRV (using extended Holter monitors), and activity (using accelerometers) every 6 months over the 2 years and evaluate if changes in wearable metrics predict changes in CMR and OGTT.

DETAILED DESCRIPTION:
Risk for hyperglycemia and insulin resistance in DMD: Individuals with DMD have multiple risk factors for abnormal glucose and insulin metabolism: frequent use of glucocorticoid (GC) medication, decreased ambulation/activity, sarcopenia, and obesity. GC use is known to increase the risk of impaired glucose tolerance (IGT) and insulin resistance (IR) in multiple populations. Decreased skeletal muscle mass and function are associated with impaired skeletal muscle insulin sensitivity and type 2 diabetes (T2D). Despite these risks, there are limited data relating glycemia and IR in this population.

This study is a critical first step in evaluating hyperglycemia in DMD and the relationship to autonomic dysfunction. Our findings will help establish screening guidelines and provide a basis for intervention studies targeting glycemia in DMD. Additionally, this study, along with other ongoing studies (Remote study: Wearable Technology to Evaluate Hyperglycemia and Heart Rate Variability in Duchenne Muscular Dystrophy) will establish wearable technology as investigational tools, for potential use in future clinical trials, in individuals with DMD and neuromuscular diseases.

Study Population: This study will include approximately 10 male participants at Vanderbilt with DMD.

DMD is an X-linked disorder affecting approximately 1/3500-6000 males and 1/50 million females. Therefore, only males will be included in this study.

Study Enrollment Period: Expected duration of the study is 6 years.

Study Visits and procedures:

Visit 1 (V1): in-person study visit

* Participants will arrive to the research clinic after an overnight fast
* Visit includes medical history, physical exam, a fasting oral glucose tolerance test (OGTT), blood will be drawn, dual-energy X-ray absorptiometry (DXA) scan, and cardiac MRI (CMR).
* Participants will wear remote monitoring devices including a continuous glucose monitor (CGM) for up to 10 days, an activity monitor (Actigraph) for up to 7 days, and a Holter (cardiac) monitor for up to 7 days.
* Participants will complete a brief diary/survey twice daily during the 7 days they are wearing the ActiGraph, Holter, and CGM. This survey will be texted or emailed to participants in the morning and evening and take approximately 5 minutes to complete. The questions are primarily related to sleep, activity, and food intake

Visit 2 (V2): remote, 6 months after Visit 1

* Participants will wear remote monitoring devices including a continuous glucose monitor (CGM) for up to 10 days, an activity monitor (Actigraph) for up to 7 days, and a Holter (cardiac) monitor for up to 7 days.
* Repeat the brief diary/survey as V1.

Visit 3 (V3): remote, 12 months after Visit 1

• Same study procedures as V2.

Visit 4 (V4): remote, 18 months after Visit 1

* Same study procedures as V2.

Visit 5 (V5): in-person study visit, approximately 24 months after Visit 1 • Same study procedures as V1.

*If the participant has completed a cardiac MRI or other study procedure for an alternate clinical or research evaluation within a month of other study procedures, the investigators may be able to use that data instead of repeating the study procedure.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

Inclusion criteria

* Male- ≥10 years
* Clinical phenotype of DMD confirmed with muscle biopsy or genotype.
* Informed consent for individuals ≥18 years
* Parent/guardian informed consent and child assent for individuals < 18 years
* Able to undergo non-sedated CMR

Exclusion Criteria

* Refusal to participate
* Diagnosis of diabetes prior to the study and/or taking insulin or other anti-diabetic drug therapy in < 4 weeks prior to treatment
* Inability to fast for 10 hours
* Use of a pacemaker, implantable cardioverter-defibrillator (ICD), or other implanted device
* Unable to comply with study procedures, in the opinion of the investigator.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — DMD is an X-linked disorder affecting approximately 1/3500-6000 males and 1/50 million females. Therefore, only males will be included in this study.
  Investigators will not obtain confirmation of biological sex and accept all participants as they self-identify.
Study Population: 10 adolescent and young adult males with DMD. DMD affects about 1/3500-6000 males and 1/50million females, therefore only male participants will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of hyperglycemia | 5 time points, each over 10 days
  number of glucose measurements ≥140mg/dL over total number of glucoses
Standard deviation of the mean R-to-R segment (SDANN) | 5 time points, each over 7 days
  correlation of rate of hyperglycemia and SDANN, which reflects heart rate variability

SECONDARY OUTCOMES:
Coefficient of variation on CGM | 5 time points, each over 10 days
  variability of glucose levels on CGM measured by coefficient of variation (COV)
Rate of significant hyperglycemia | 5 time points, each over 10 days
  number of glucose measurements ≥200mg/dL over total number of glucoses
Activity level | 5 time points, each over 7 days
  Time spent in sedentary, low intensity, and moderate to vigorous physical activity
Standard deviation of normal R to R intervals (SDNN) | 5 time points, each over 7 days
  correlation of rate of hyperglycemia and SDNN
Late gadolinium enhancement (LGE) | 2 time points: initially and approximately 2 years later
  correlation of change in SDANN from 0 to 24 months with change in percent LVEF on cardiac MRI from 0 to 24 months
Left ventricular ejection fraction (LVEF) | 2 time points: initially and approximately 2 years later
  correlation of change in SDANN from 0 to 24 months with change in percent LVEF on cardiac MRI from 0 to 24 months
Insulin sensitivity | 2 time points: initially and approximately 2 years later
  correlation between change in rate of hyperglycemia from 0 to 24 months (CGM) with change in insulin sensitivity from 0 to 24 months (oral glucose tolerance test)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Tamaroff, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No